CLINICAL TRIAL: NCT02455570
Title: Global Assessment of Endoscopic Ultrasound Performance Skills - a New Tool to Measure the Learning Curve and Technical Skills of Endosonografists
Brief Title: Global Assessment of Endoscopic Ultrasound Performance Skills
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Per Hedenström, Dr, Sahlgrenska University Hospital
Other Study IDs: Dnr 721-13
Record Dates: First submitted 2015-05-22; First posted 2015-05-28 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: E01.370.350.850.280; I02.399; J01.897.608; N06.850.135.060.075.399; F02.784.629.529.274
Keywords: Endoscopic Ultrasound; Quality Management; Education and training; Safety; Learning curve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Endoscopic ultrasound (EUS) is a mini-invasive diagnostic procedure in the work-up of various suspicious malignancies. The learning curve of EUS is regarded long but so far the literature of this topic is minimal. Few studies have been published and there are no standardized or validated methods to perform a systematic assessment of endosonographists in training. This study is an observational study dealing with the matter of assessing endosonographists in training.

DETAILED DESCRIPTION:
Sahlgrenska Univeristy Hospital is tertiary university endoscopy center. At our endoscopy unit physicians/endoscopists train EUS under the supervision of an experienced endosonographist. Endosonographists examining patients referred for a routine, clinical EUS at the Sahlgrenska Univeristy hospital are candidates for being study subjects. Patients will not be examined by the study endosonographists if supervision is lacking.

External, collaborating centers will be invited to participte in the study given that the study inclusion criteria and ethical standard will be ensured.

The investigators of this study have developped a score sheet for the assessment of endosonographists in training to be used in a standard clinical setting. The score sheet is to be used by both the endosonographist in training (performer) for self-assessment and by the supervisor (observer) for assessment of the performer.

First, background data of the performer is recorded (pervious endoscopy experience etc). Then the performer starts the examination under the guidance of the observer. The observer performs continuous evaluation and assessment of the performer according to the skill parameters (N=5) of the Observer score sheet. Each parameter is ranked on a 1-5 scale (1=non-satisfactory performance, 5= excellent performance). Finally the observer is taking over, reevaluates the findings of the performer and finishes the examination.

After the examination the performer fullfills the Performer score sheet. Finally, both the performer and the observer record their preliminary diagosis of the lesion examined.

Adverse events and complications are recorded.

A follow-up of the medical records of the patient is performed 8 weeks after the EUS-examiantion with respect to the final diagnosis of the lesion of interest. The reference standard is set to best available combination of surgery, pathology and imaging reports. The performer´s assessment of the diagnosis is the categorized as CORRECT or FALSE. A correct diagnosis equals 3 Points and a false diagnosis equals 0 Points.

Results in terms of the total and mean score of all perfomers is calculated and collected in a study database. Feasibility of the study assessment sheet is evaluated. Statistical analysis of categorical data is finally applied for evaluating the results with respect to the progress and learning curve of the study participants.

ELIGIBILITY:
Inclusion Criteria:

* EUS-examination with or without sampling performed for clinical reasons at one of the participating centers
* The EUS-examination is to be performed by a physician in training as endosonographist OR a physician with a completed training as endosonographist
* The EUS-examination is to be supervised by an experienced endosonographist
* Oral and written consent of the patients examined (age>18 years)

Exclusion Criteria:

* Physicians in EUS-traning without adequate supervision
* Experimental or therapeutic EUS outside the clinical setting

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Endosonographists in traning under experienced supervision at tertiary endoscopy centers.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-08; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
EUS performance | Imediate
  The assessment and scoring of the endosonographist in training (Performer) is performed during the EUS-examiantion itself by the supervisor (Observer) in real-time. The total score is a compound of five parameters assessed each on a 1-5 scale (1=non-satisfactory performance, 5=excellent performance). A study unique assessment sheet is developped.

SECONDARY OUTCOMES:
EUS diagnosis | 2 months
  The performer states his/her preliminary diagnosis of the lesion examined by EUS based on his/her findings. The correct diagnosis of the examined lesion is reviewed and recorded from surgery/pathology/imaging reports of the medical files in each individual case at a time frame of 8 weeks after EUS. The preliminary diagnosis stated by the performer is then categorized as CORRECT or FALSE.
Safety and complications | <48 hours
  Adverse events and complications occuring during the procedure or within 48 hours with a potential causal relation to the EUS-examination is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Riadh Sadik, Ass prof, Principal Investigator — Sahlgrenska University Hospital, Gothenburg
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Wani S, Cote GA, Keswani R, Mullady D, Azar R, Murad F, Edmundowicz S, Komanduri S, McHenry L, Al-Haddad MA, Hall M, Hovis CE, Hollander TG, Early D. Learning curves for EUS by using cumulative sum analysis: implications for American Society for Gastrointestinal Endoscopy recommendations for training. Gastrointest Endosc. 2013 Apr;77(4):558-65. doi: 10.1016/j.gie.2012.10.012. Epub 2012 Dec 20. PMID 23260317
- [Derived] Hedenstrom P, Marasco G, Eusebi LH, Lindkvist B, Sadik R. GAPS-EUS: a new and reliable tool for the assessment of basic skills and performance in EUS among endosonography trainees. BMJ Open Gastroenterol. 2021 Jun;8(1):e000660. doi: 10.1136/bmjgast-2021-000660. PMID 34108134